CLINICAL TRIAL: NCT05776290
Title: Evaluation of the Efficacy of a Hyaluronic Acid Gel in Relieving Post-Implantation Pain: A Split-Mouth Randomized Controlled Trial
Brief Title: The Effect of Hyaluronic Acid Gel on Relieving Post-Implantation Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OralMed-01-2023
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Implant Complication
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid injection (Experimental): The hyaluronic acid will be injected into the implant socket before implantation.
  Interventions: Biological: Hyaluronic Acid
- Traditional treatment (No Intervention): The socket will be prepared in the normal manner without being injected with any material.

INTERVENTIONS:
Biological: Hyaluronic Acid — This material will be injected into the prepared impact socket prior to inserting the implant. This injection will be done inside the socket as well as on the periphery of the socket.
  Arms: Hyaluronic acid injection

SUMMARY:
Few previous studies have employed HA in the implant socket; instead, the majority have applied it topically to the area around dental implants after they have been placed. The application was done after suturing in these investigations. Therefore, the goal of the current study was to inject HA into the implant socket and onto the alveolar bone prior to implant insertion and suturing in order to preserve the HA for an extended period of time.

This study aims to use a visual analog scale (VAS) on the first, third, and tenth days following the surgical intervention to assess the efficacy of employing HA in dental implants in terms of pain reduction that may accompany dental implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* bilateral tooth loss with a sufficient amount of bone volume
* no general problems
* good oral health
* age between 20 and 60 years

Exclusion Criteria:

* the use of immunosuppressive drugs and corticosteroids for long periods
* the existence of serious systemic disorders
* contraindications for local anesthesia or oral surgery
* pregnant women and nursing mothers
* patients receiving chemotherapy or radiation
* alcoholics and heavy smokers.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Change in the Perception of pain | First assessment: at 24 hours following the surgical procedure. Second assessment: at 72 hours following the surgical intervention. Third assessment will be made on the tenth day following the surgical intervention
  This will be measured using a numeric rating scale. Patients will be asked to indicate the level of pain they perceive on a scale from 1 to 10. The intensity of pain is going to be classified according to the following categories: 0 = no pain, 1-3 = mild pain, 3-6 = moderate pain, and 6-10 = severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Al-Khateeb, DDS MSc, Principal Investigator — PhD student at the Department of Oral Medicine
Locations (1):
- Department of Oral Medicine, Faculty of Dentistry, University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
Datasets and the underlying worksheets are available upon reasonable request from the corresponding author once the paper has been published.